CLINICAL TRIAL: NCT03251872
Title: Olaparib for Pulmonary Arterial Hypertension: a Pilot Clinical Study
Brief Title: Olaparib for PAH: a Pilot Study
Acronym: OPTION-p
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: OPTION pilot trial merged with the new NCT03782818 - OPTION multicenter trial
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Steeve Provencher, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-21658
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH; poly (ADP-ribose) polymerases inhibition; PARP-1 inhibition; DNA damage; Early-phase clinical trial pilot study; Olaparib; Safety and efficacy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: The design is open-label. A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of medication. Patients will be given progressive doses of olaparib up to 400mg BID for 16 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: Olaparib (Experimental): Olaparib up to 400 mg BID (100 to 400 mg) for 16 weeks
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib tablets
  Other Names: Lynparza

SUMMARY:
The main OBJECTIVE of this proposal is to extend our preclinical findings on the role of DNA damage and poly(ADP-ribose) polymerases (PARP) inhibition as a therapy for a devastating disease, pulmonary arterial hypertension (PAH), to early-phase clinical trials. We, and others, have published strong evidence that DNA damage accounts for disease progression in PAH and showed that PARP1 inhibition can reverse PAH in several animal models1. Interestingly, PARP1 inhibition is also cardioprotective. Olaparib, an orally available PARP1 inhibitor, can reverse cancer growth in animals and humans with a good safety profile, and is now approved for the treatment of ovarian cancer in Canada, Europe and the USA. The time is thus right to translate our findings in human PAH. The industry-sponsored clinical research on PARP1 inhibitor is currently entirely cancer-oriented. Nonetheless, AstraZeneca Canada accepted to support an early phase clinical trial through in-kind contribution, but the support from foundations and federal agencies is critical to catalyze early-stage development of PARP1 inhibitors for other indications, especially for orphan diseases. A CIHR Project Scheme grant will thus be submitted on September 15 2017, proposing a Phase 1, followed by a Phase 2 trial that will be conducted in recognized PAH programs throughout Canada. At this stage, however, we propose a pilot study to assess the feasibility of the proposed trials in the PAH population. The overall HYPOTHESIS is that PARP1 inhibition with olaparib is a safe and effective therapy for PAH.

The primary objective of the study is to confirm feasibility, to support the safety of using olaparib in PAH patients, and precise the sample size of the coming Phase 1B trial. The feasibility of the comprehensive patient phenotyping that will be proposed within the phase 1B trial will thus be assessed, in addition to adverse events and efficacy signals.

***OPTION pilot trial was merged with the new OPTION multicenter trial (NCT03782818)***

DETAILED DESCRIPTION:
BACKGROUND PAH is a progressive and multifactorial condition characterized by the chronic elevation of pulmonary artery (PA) pressure leading to RV failure. In spite of currently approved therapies, patients with PAH have poor quality of life and the 3-year survival of idiopathic PAH remains ~55%. The identification and characterization of new therapeutic targets is thus an urgent need.

In recent years, it has become increasingly appreciated that, as in cancer cells, PAH-PA smooth muscle cells (PASMCs) are exposed to stressful conditions, jeopardizing their survival. To deal with these insults, these cells have developed complementary pathways, allowing them to survive and proliferate and leading to intense remodelling of distal PA. Central to these strategies are the activation of the DNA repair machinery. Survival of these cells is associated with an over-efficient activation of PAPR1, a predominant mechanism involved in DNA repair, and pharmacological inhibition of PARP1 reverses PAH in human cells and clinically relevant animal models.

Recently, Olaparib, an orally available PARP1 inhibitor, was shown to be safe, well tolerated and effective in treating cancers and was approved for the treatment of ovarian cancer.

OLAPARIB IN PAH: A PILOT STUDY The study population will include 6 well-characterized PAH patients that have been stable for >4 months on standard PAH-therapies, as per guidelines.

The primary objective of the study is to confirm the feasibility for a future early stage clinical trial and provide early evidence that Olaparib may be effective in PAH.

Exploratory efficacy end-point: The exploratory efficacy endpoint will be the change in pulmonary vascular resistance (PVR) at week 16. Other exploratory efficacy end-points will include changes in: 1) additional haemodynamic data by catheterization; 2) 6-min walk distance (6MWD); 3) RV volumes and mass (cardiac MRI) in eligible patients; 4) WHO functional class; 5) NT-proBNP levels; 6) Quality of life assessed using the CAMPHOR questionnaire.

Study design: This is a standard-design, dose-escalating pilot study. In line with most pilot and safety studies, the design is open-label. A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of medication. Patients will be given progressive doses of olaparib up to 400mg BID for 16 weeks. Patients will be regularly followed. At baseline and week 16, a cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function.

Toxicity monitoring/withdrawal: Based on experience to date with olaparib, doses up to 400mg BID should be tolerated. Subjects may experience mild side effects or other events that the investigator may consider related to study drug but not of sufficient clinical significance to warrant withdrawal from treatment. At the investigators' discretion, olaparib may be managed by dose reduction. If the lower dose is not tolerated, the patient will be withdrawn from the study. Subjects who require a dose reduction should be maintained at the reduced dose level through to the end of the 16-week treatment period. Adverse events will be submitted to our ethics committees.

Analysis: This pilot study is not meant to prove efficacy. As a result, power calculations were not determined. The safety and exploratory endpoint analysis will be only descriptive. Nonetheless, it is hoped that olaparib will be associated with hemodynamic improvements, giving precision about the dose to be tested and sample size calculation for subsequent studies. Thus, there is a need for assessment of the exploratory efficacy endpoints. These analyses will be based on the per protocol set (all treated patients who did not violate the protocol in a way that might influence the evaluation of the effect of the study drug on the primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* 1) adults (18-75 yrs) with PAH of idiopathic/ hereditary/drug or toxin-induced origin or associated with connective tissue diseases; 2) mean PA pressure ≥25mmHg, PA wedge pressure ≤15mmHg, PVR >480 dyn.s.cm-5 and absence of acute vasoreactivity (we expect PARP1 inhibition will be most effective in patients with significant PA remodelling); 3) WHO functional class II or III; 4) clinically stable with unchanged vasoactive therapy for ≥4 months; 5) two 6MWD of 150-550m and within ±15% of each other (the latter being used as baseline value); 6) a negative serum pregnancy test prior to receiving the first dose of study treatment and willing to use adequate contraception from enrolment through 3 months after the last dose of study treatment for patients of childbearing potential

Exclusion Criteria:

* 1) other types of pulmonary hypertension; 2) significant restrictive (total lung capacity <60% predicted) or obstructive (FEV1/FVC<60% after a bronchodilator) lung disease; 3) systolic blood pressure <90 mmHg; 4) acute RV failure within the last 3 months; 5) received any investigational drug within 30 days; 6) BMI <18 or >40 kg/m2; 7) cardiopulmonary rehabilitation program planned or started ≤12 weeks prior to Day 1; 8) presence of ≥3 risk factors for heart failure with preserved ejection fraction (BMI >30 kg/m2, diabetes mellitus, hypertension or coronary artery disease); 9) organ dysfunction other than RV failure; 10) anticipated survival <1 year due to concomitant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR) at week 16 | 16 weeks
  At baseline and week 16, a cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function

OTHER OUTCOMES:
Additional haemodynamic data by catheterization | At baseline and week 16
  A cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function
6-min walk distance (6MWD) | At baseline and week 16
  The six-minute walk test (6MWT) measures the distance (6MWD) that a person can quickly walk on a flat, hard surface in 6 min.
RV volumes and mass (cardiac MRI) | At baseline and week 16
  A cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function
WHO functional class | At baseline and week 16
  Assesses the severity of the disease using a range of clinical assessments, exercise tests, biochemical markers, and echocardiographic and haemodynamic assessments. The clinical assessment of the patient has a pivotal role in the choice of the initial treatment, the evaluation of the response to therapy, and the possible escalation of therapy if needed. The clinical severity of PAH is classified by the World Health Organization (WHO) according to a system that grades PAH severity according to the functional status of the patient. The grades range from Functional Class (FC) I, where the patient's disease does not affect their day-to-day activities, to FC IV, where patients are severely functionally impaired, even at rest. This functional classification system links symptoms with activity limitations, and allows clinicians to quickly predict disease progression and prognosis, as well as the need for specific treatment regimens, irrespective of the underlying aetiology of PAH.
NT-proBNP levels | At baseline and week 16
  Blood test. B-type natriuretic peptide (brain natriuretic peptide: BNP) is a small, ringed peptide secreted by the heart to regulate blood pressure and fluid balance. This peptide is stored in and secreted predominantly from membrane granules in the heart ventricles in a pro form (proBNP). Once released from the heart in response to ventricle volume expansion or pressure overload, the N-terminal (NT) piece of 76 amino acids (NT-proBNP) is rapidly cleaved by the enzymes corin and furin to release the active 32-amino acid peptide (BNP). Both BNP and NT-proBNP are markers of atrial and ventricular distension due to increased intracardiac pressure.
Quality of life - Clinical deterioration | At baseline and week 16
  Assessed using the CAMPHOR questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — IUCPQ-UL; Sébastien Bonnet, PhD, FAHA, Principal Investigator — IUCPQ-UL
Locations (1):
- IUCPQ-UL, Québec, Quebec, Canada

REFERENCES:
- [Background] Chen PI, Cao A, Miyagawa K, Tojais NF, Hennigs JK, Li CG, Sweeney NM, Inglis AS, Wang L, Li D, Ye M, Feldman BJ, Rabinovitch M. Amphetamines promote mitochondrial dysfunction and DNA damage in pulmonary hypertension. JCI Insight. 2017 Jan 26;2(2):e90427. doi: 10.1172/jci.insight.90427. PMID 28138562
- [Background] de Jesus Perez VA, Yuan K, Lyuksyutova MA, Dewey F, Orcholski ME, Shuffle EM, Mathur M, Yancy L Jr, Rojas V, Li CG, Cao A, Alastalo TP, Khazeni N, Cimprich KA, Butte AJ, Ashley E, Zamanian RT. Whole-exome sequencing reveals TopBP1 as a novel gene in idiopathic pulmonary arterial hypertension. Am J Respir Crit Care Med. 2014 May 15;189(10):1260-72. doi: 10.1164/rccm.201310-1749OC. PMID 24702692
- [Background] Dedes KJ, Wetterskog D, Mendes-Pereira AM, Natrajan R, Lambros MB, Geyer FC, Vatcheva R, Savage K, Mackay A, Lord CJ, Ashworth A, Reis-Filho JS. PTEN deficiency in endometrioid endometrial adenocarcinomas predicts sensitivity to PARP inhibitors. Sci Transl Med. 2010 Oct 13;2(53):53ra75. doi: 10.1126/scitranslmed.3001538. PMID 20944090
- [Background] Federici C, Drake KM, Rigelsky CM, McNelly LN, Meade SL, Comhair SA, Erzurum SC, Aldred MA. Increased Mutagen Sensitivity and DNA Damage in Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2015 Jul 15;192(2):219-28. doi: 10.1164/rccm.201411-2128OC. PMID 25918951
- [Background] Happe CM, Szulcek R, Voelkel NF, Bogaard HJ. Reconciling paradigms of abnormal pulmonary blood flow and quasi-malignant cellular alterations in pulmonary arterial hypertension. Vascul Pharmacol. 2016 Aug;83:17-25. doi: 10.1016/j.vph.2016.01.004. Epub 2016 Jan 22. PMID 26804008
- [Background] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Background] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Macpherson E, Watkins C, Carmichael J, Matulonis U. Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med. 2012 Apr 12;366(15):1382-92. doi: 10.1056/NEJMoa1105535. Epub 2012 Mar 27. PMID 22452356
- [Background] Li M, Vattulainen S, Aho J, Orcholski M, Rojas V, Yuan K, Helenius M, Taimen P, Myllykangas S, De Jesus Perez V, Koskenvuo JW, Alastalo TP. Loss of bone morphogenetic protein receptor 2 is associated with abnormal DNA repair in pulmonary arterial hypertension. Am J Respir Cell Mol Biol. 2014 Jun;50(6):1118-28. doi: 10.1165/rcmb.2013-0349OC. PMID 24433082
- [Background] Meloche J, Le Guen M, Potus F, Vinck J, Ranchoux B, Johnson I, Antigny F, Tremblay E, Breuils-Bonnet S, Perros F, Provencher S, Bonnet S. miR-223 reverses experimental pulmonary arterial hypertension. Am J Physiol Cell Physiol. 2015 Sep 15;309(6):C363-72. doi: 10.1152/ajpcell.00149.2015. Epub 2015 Jun 17. PMID 26084306
- [Background] Meloche J, Pflieger A, Vaillancourt M, Paulin R, Potus F, Zervopoulos S, Graydon C, Courboulin A, Breuils-Bonnet S, Tremblay E, Couture C, Michelakis ED, Provencher S, Bonnet S. Role for DNA damage signaling in pulmonary arterial hypertension. Circulation. 2014 Feb 18;129(7):786-97. doi: 10.1161/CIRCULATIONAHA.113.006167. Epub 2013 Nov 22. PMID 24270264
- [Background] Moudry P, Watanabe K, Wolanin KM, Bartkova J, Wassing IE, Watanabe S, Strauss R, Troelsgaard Pedersen R, Oestergaard VH, Lisby M, Andujar-Sanchez M, Maya-Mendoza A, Esashi F, Lukas J, Bartek J. TOPBP1 regulates RAD51 phosphorylation and chromatin loading and determines PARP inhibitor sensitivity. J Cell Biol. 2016 Feb 1;212(3):281-8. doi: 10.1083/jcb.201507042. Epub 2016 Jan 25. PMID 26811421
- [Background] Park ES, Kang DH, Kang JC, Jang YC, Lee MJ, Chung HJ, Yi KY, Kim DE, Kim B, Shin HS. Cardioprotective effect of KR-33889, a novel PARP inhibitor, against oxidative stress-induced apoptosis in H9c2 cells and isolated rat hearts. Arch Pharm Res. 2017 May;40(5):640-654. doi: 10.1007/s12272-017-0912-3. Epub 2017 Apr 4. PMID 28378219
- [Background] Rabinovitch M, Guignabert C, Humbert M, Nicolls MR. Inflammation and immunity in the pathogenesis of pulmonary arterial hypertension. Circ Res. 2014 Jun 20;115(1):165-75. doi: 10.1161/CIRCRESAHA.113.301141. PMID 24951765
- [Background] Ramsey BW, Nepom GT, Lonial S. Academic, Foundation, and Industry Collaboration in Finding New Therapies. N Engl J Med. 2017 May 4;376(18):1762-1769. doi: 10.1056/NEJMra1612575. No abstract available. PMID 28467868
- [Background] Ranchoux B, Meloche J, Paulin R, Boucherat O, Provencher S, Bonnet S. DNA Damage and Pulmonary Hypertension. Int J Mol Sci. 2016 Jun 22;17(6):990. doi: 10.3390/ijms17060990. PMID 27338373
- [Background] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- See also: OPTION pilot trial merged to a new multicenter trial (OPTION multicenter - NTC03782818) — https://clinicaltrials.gov/ct2/show/NCT03782818?term=NCT03782818&draw=2&rank=1